CLINICAL TRIAL: NCT02051803
Title: Distress Tolerance Treatment for Weight Concern in Smoking Cessation Among Women
Brief Title: Women Engaging in Quitting Smoking Together (WE QUIT)
Acronym: WE QUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1303-003; K23DA035288 (NIH)
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; women
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Distress Tolerance Treatment for Weight Concern (DT-W) (Experimental): DT-W is delivered over a 9 week period with 1 1-hr individual session during week 1, 8 weekly 1.5-hr group counseling sessions during weeks 2-9, and 1 20-minute individual telephone session during week 4. Session content includes distress tolerance intervention for weight concern plus standard behavioral smoking cessation treatment. Participants also receive 8 weeks of nicotine patch.
  Interventions: Behavioral: Distress Tolerance Treatment for Weight Concern (DT-W)
- Health Education (HE) (Active Comparator): HE is delivered over a 9 week period with 1 1-hr individual session during week 1, 8 weekly 1.5-hr group counseling sessions during weeks 2-9, and 1 20-minute individual telephone session during week 4. Session content includes smoking health education program plus standard behavioral smoking cessation treatment. Participants also receive 8 weeks of nicotine patch.
  Interventions: Behavioral: Health Education (HE)

INTERVENTIONS:
Behavioral: Distress Tolerance Treatment for Weight Concern (DT-W)
  Arms: Distress Tolerance Treatment for Weight Concern (DT-W)
Behavioral: Health Education (HE)
  Arms: Health Education (HE)

SUMMARY:
The long-term goal of this program of research is to develop and disseminate an efficacious intervention for weight concern that will significantly increase smoking cessation rates among women. The overall objective of this project is to develop this intervention and modify it based on piloting and feedback to ensure its feasibility and acceptability. These objectives will be accomplished by pursuing the following specific aim: 1) develop a group-based distress tolerance treatment for weight concern (DT-W) in female smokers and a comparison health education (HE) program and pilot both treatments with three groups of 10 (total N = 30) female weight-concerned smokers (2 DT-W groups, 1 HE group).

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 to 65 years of age
* smoke 10 or more cigarettes per day
* daily smoker for at least the past year
* report motivation to quit smoking in the next month of at least 5 on a 10 point scale
* report concern of at least 50 on at least one of two 100 point scales assessing weight concern
* able to travel to study location for study appointments

Exclusion Criteria:

* current use of other smoking cessation or weight loss therapies
* current use of other tobacco products at least weekly
* current diagnosis of depression
* diagnosis or treatment for non-nicotine substance use disorder with substance use during the past 6 months
* lifetime diagnosis or treatment of eating disorder, bipolar disorder, schizophrenia, or schizoaffective disorder
* current use of psychotropic medication except antidepressants
* score above established cut-offs on self-report screening measures of depressive symptomology, eating disorder symptomology, alcohol use disorder, or drug use disorder
* current suicidality or homicidality
* medical condition that is a contraindication for the use of transdermal nicotine patch
* lives at same address as current or past participant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence from smoking | 6 months from smoking quit date
  We will compare the percentage of participants in each treatment group who report abstinence from smoking for the 7 days prior to each follow-up assessment (1-, 3-, and 6-months post-quit date).

CONTACTS AND LOCATIONS:
Overall Officials: Erika L. Bloom, Ph.D., Principal Investigator — Butler Hospital and Rhode Island Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States